CLINICAL TRIAL: NCT06370624
Title: Quantitative Assessment of Cerebral Vascular Reactivity by Resting Functional Magnetic Resonance Imaging of Infants With Hypoxic Ischemic Encephalopathy After Hypothermia Treatment: Diagnostic and Prognostic Implications.
Brief Title: PEDI-REAVASC Resonance Imaging of Infants With Hypoxic Ischemic Encephalopathy After Hypothermia Treatment.
Acronym: PEDI-REAVASC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022/03OCT/360
Record Dates: First submitted 2024-04-09; First posted 2024-04-17 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Encephalopathy, Hypoxic-Ischemic
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: One group will be followed - with both the standard of care continuous EEG monitoring and near infrared spectroscopy (NIRS) & the MRI-scan performed at the same time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Newborns (Experimental)
  Interventions: Diagnostic Test: MRI-scan

INTERVENTIONS:
Diagnostic Test: MRI-scan — IRM-scan at rest under neonatologist monitoring.

SUMMARY:
This study is a prospective, observational, single-center study to assess the correlation between rs-fMRI measures and clinical measures of standard MRI, NIRS, EEG and clinical scores.

The target population was neonates with HIE referred to MRI after hypothermia treatment, which was initiated within 6 hours of birth, continued for 72 hours and followed by a slow rewarming period of 6-12 hours.

A one-year clinical and imaging follow-up is planned. As the aim of the present study is to assess the predictiveness of the outcome one year after the HIE event, no follow-up is planned.

ELIGIBILITY:
Inclusion Criteria:

Newborns at 36 weeks gestation or more, with HIE treated with therapeutic hypothermia will be prospectively included.

Exclusion Criteria:

* Lack of parental consent
* Congenital anomalies that make hypothermia treatment not indicated
* Coagulopathy with active bleeding

Ages: 1 Hour to 14 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
quantifying cerebrovascular reactivity (CVR) by resting-state functional MRI (r-fMRI) in infants with moderate to severe hypoxic-ischaemic encephalopathy (HIE) | at birth, directly after hypothermia and at 1 year of baby's life
  Correlation between RCV mapping EEG/MRI

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Onofrj, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint Luc, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No